CLINICAL TRIAL: NCT02197065
Title: The Post-Operative Statin for Thromboprophylaxis & Cardiovascular Outcomes Protection (POST-OP) Pilot Trial
Brief Title: Pilot Study of Atorvastatin for Orthopedic Surgery Patients
Acronym: POST-OP Pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Weill Medical College of Cornell University (Other); Washington University School of Medicine (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EPAR4398; UL1TR000457-06 (NIH)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-04

CONDITIONS: Hip Fracture; Myocardial Ischemia; Inflammation
Keywords: hip fracture; myocardial ischemia; statin; surgery; troponin; complication; arthroplasty; hip; knee; orthopedic; atorvastatin; cardiovascular
MeSH Terms: conditions — Hip Fractures; Myocardial Ischemia; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin 40mg daily starting at least 4 hours prior to hip fracture surgery, or 4 days prior to hip or knee arthroplasty, and continued until postoperative day 45.
  Interventions: Drug: Atorvastatin
- Sugar pill (Placebo Comparator): Sugar pill (placebo) daily starting at least 4 hours prior to hip fracture surgery, or 4 days prior to hip or knee arthroplasty, and continued until postoperative day 45.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin or placebo will be started at least 4 hours prior to surgery, and continued nightly until postoperative day 45
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo
  Arms: Sugar pill

SUMMARY:
Up to 35% of hip fracture patients have been shown to experience heart injury after surgery, and as many as 10% have a heart attack or die in the three months after surgery. Hip and knee arthroplasty patients are also at risk of cardiovascular complications. Patients who have these complications have higher levels of inflammation postoperatively. Statins (such as atorvastatin/Lipitor) lower cholesterol and also lessen inflammation. Both of these effects are important in preventing heart attacks. Statins have been shown to reduce the risk of heart attacks in non-surgical patients, and to protect from heart attacks in patients having heart surgery. Whether statins can prevent heart attacks in orthopedic patients is not known.

In this pilot study the investigators will treat 30 orthopedic surgery patients (hip fracture, hip or knee arthroplasty) with either atorvastatin or placebo (a capsule with no study drug). Patients will start the study drug prior to surgery and take it for 45 days after surgery. Neither the doctors nor the patients will know whether they are taking atorvastatin or placebo. The investigators will look for evidence of inflammation and heart injury after surgery. The investigators hypothesize that atorvastatin will lessen the degree of postoperative inflammation found in these patients. In this study, the investigators will use a very sensitive test of heart injury that can detect problems even when patients have no symptoms. The investigators hypothesize that this test will demonstrate silent heart injury in over 50% of the hip fracture patients and over 30% of arthroplasty patients in our study.

The results of this trial will help us to develop a larger study in 1000 hip fracture and joint replacement patients to determine whether atorvastatin protects orthopedic surgery patients from heart injury and other complications of surgery.

DETAILED DESCRIPTION:
* Thirty statin-naïve patients ≥ 65 years of age admitted to New York Presbyterian Hospital or Hospital for Special Surgery with an acute hip fracture, or for elective hip or knee arthroplasty will be randomized in a 1:1 ratio to atorvastatin 40 mg daily or matching placebo.
* Atorvastatin will be initiated at least 4 hours prior to hip fracture surgery, or 4 days prior to arthroplasty, and will be continued until postoperative day (POD) 45.
* Patients will be assessed daily in the hospital for adverse events.
* Patients will be contacted by telephone weekly for four weeks after surgery and again on POD 45 and POD 90.
* Patients will mail back study medication bottles on POD 45 for pill counts to assess compliance.
* High sensitivity cardiac troponin I (hs-cTnI) will be measured pre-operatively (prior to atorvastatin therapy) and on POD 2.
* High sensitivity C-reactive protein (hs-CRP), and a panel of cytokines (IL-1β, IL-2, IL-2r, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-17, tumor necrosis factor (TNF)-α, interferon (IFN)-γ, and soluble (s)CD-40L) will be measured preoperatively and on POD 2.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture or elective hip or knee arthroplasty
* Age 65 years or older
* Life expectancy > 3 months

Exclusion Criteria:

* Pathological hip fracture due to cancer
* Currently taking a statin, or took a statin within the last 30 days
* Previous statin intolerance
* Acute myocardial infarction or unstable angina
* History of myocardial infarction, acute coronary syndrome, angina, coronary/arterial re-vascularization
* Hip fracture patients with peripheral arterial disease
* Hip fracture patients with history of stroke or transient ischemic attack.
* Muscle disorder
* Serious liver disease or alanine aminotransferase > 3x upper limit of normal
* Serious renal disease (creatinine clearance <30cc/min)
* Treatment with HIV protease inhibitor or Hepatitis C protease inhibitor
* Treatment with erythromycin, clarithromycin, niacin or azole antifungal agent
* Pregnant, planning to become pregnant, or breastfeeding

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne R Bass, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (2):
- United States (2):
  - Hospital for Special Surgery, New York, New York
  - New York Presbyterian Hospital (Cornell), New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bass AR, Szymonifka JD, Rondina MT, Bogardus M, Scott MG, Woller SC, Stevens SM, Eby C, Merritt K, Valle AGD, Moskowitz G, Flores E, Gage BF. Postoperative Myocardial Injury and Inflammation Is Not Blunted by a Trial of Atorvastatin in Orthopedic Surgery Patients. HSS J. 2018 Feb;14(1):67-76. doi: 10.1007/s11420-017-9577-1. Epub 2017 Oct 13. PMID 29398998

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: Sugar pill (placebo) daily starting at least 4 hours prior to hip fracture surgery, or 4 days prior to hip or knee arthroplasty, and continued until postoperative day 45.
  Placebo
Period: Overall Study
Arm/Group | Atorvastatin | Sugar Pill
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Sugar Pill | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [67 to 76] | 75 [72 to 84] | 73 [70 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Orthopedic procedure [Count of Participants; unit: Participants]
  Knee arthroplasty | 2 | 4 | 6
  Hip arthroplasty | 6 | 4 | 10
  Hip fracture repair | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of All Enrolled Patients With a Peri-operative Rise in High-sensitivity Cardiac Troponin I
Description: The percentage of orthopedic patients with a ≥ 10 pg/mL rise in high-sensitivity cardiac troponin I (hs-cTnI) from baseline pre-operatively to post-operative day (POD)2
Time Frame: change from preoperative to postoperative day 2
Population: 20 orthopedic surgery patients.
Measure: Number; unit: percentage of patients
Groups:
- All Patients: All patients in the study
Arm/Group | All Patients
Number analyzed (Participants) | 20
percentage of patients | 20
Statistical Analysis 1: Comparison: All Patients; This was a pilot feasibility study and we were only powered to determine the frequency of troponin elevation in the entire study population, not to compare the frequency of a rise in troponin in the two study arms. Thus Aim 1 applies to the entire study cohort; Test type: Other; Proportion = 0.2

2. Primary Outcome: Peri-operative Rise in High Sensitivity C-reactive Protein (Hs-CRP)
Description: The change in the level of hs-CRP from baseline to POD2 in 20 orthopedic patients randomized (1:1) to atorvastatin 40mg versus placebo.
Time Frame: Change from preoperative to post-operative day 2
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 10 | 10
mg/L | 98.95 [63.8 to 151.4] | 85.95 [52.85 to 124.9]
Statistical Analysis 1: Comparison: Atorvastatin vs Sugar Pill; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 13

3. Secondary Outcome: Peri-operative Rise in Interleukin-6 (IL-6) Levels
Description: The change in the level of IL-6 from baseline to POD2 in 16 arthroplasty patients randomized (1:1) to atorvastatin 40mg versus placebo.
Time Frame: Change from preoperative to postoperative day 2
Population: 16 arthroplasty patients
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Atorvastatin: Atorvastatin 40mg daily starting 4 days prior to hip or knee arthroplasty, and continued until postoperative day 45.
- Sugar Pill: Sugar pill (placebo) daily starting 4 days prior to hip or knee arthroplasty, and continued until postoperative day 45.
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 8 | 8
pg/mL | 1.28 [0.09 to 1.58] | 0.98 [0.53 to 1.45]
Statistical Analysis 1: Comparison: Atorvastatin vs Sugar Pill; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.3

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Atorvastatin | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/10
Other Adverse Events (participants affected / at risk) | 3/10 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=10) | Sugar Pill (N=10)
deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) — calf vein
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
bacteremia (Infections and infestations) | 0 (0) | 1 (1)
delirium (Nervous system disorders) | 0 (0) | 1 (1)
alcohol withdrawal (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
fluid overload (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=10) | Sugar Pill (N=10)
Infection (Infections and infestations) | 3 (4) | 2 (2)
delirium (Nervous system disorders) | 2 (2) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size: recruitment was made difficult by comorbidities in hip fracture patients that limited participation, the reluctance of arthroplasty patients to enroll in an interventional trial, and statin use in 40% of the target population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No